CLINICAL TRIAL: NCT00177658
Title: NCCLS Interpretive Criteria for Salmonella
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB # 0602124 (Old #0303110)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Salmonella Infection
Keywords: Salmonella
MeSH Terms: conditions — Salmonella Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To determine the clinical significance of gene mutations encoding antibiotic resistance, but not expressed as clinical resistance, in Salmonella bacteria

DETAILED DESCRIPTION:
Observational study. Physicians in foreign countries caring for patients with Salmonella meningitis or bloodstream infections will collect data on the patients they care for and send this data and an isolate of the organism causing the infection to the University of Pittsburgh.

ELIGIBILITY:
Inclusion Criteria:

* salmonella positive isolate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: isolates with salmonella
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States